CLINICAL TRIAL: NCT05289934
Title: Effects of Recorded Music on Clinical and Electroencephalography (EEG) Seizure Activity
Brief Title: Effects of Recorded Music on Clinical and EEG Seizure Activity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00260509
Record Dates: First submitted 2022-03-10; First posted 2022-03-22 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Epilepsy
Keywords: Epilepsy; Electroencephalography (EEG); Music
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Intervention Model Description: The children will listen to Mozart K.448 (1st movement) and instrumental age-appropriate songs with 10 minutes wash out in between, each lasting up to 9 minutes in the daytime (between 1-5 pm). The order of music stimuli will be randomly played in 2 to 7 days during the Epilepsy Monitoring Units (EMU) stay. Standard clinical care recording continuous video electroencephalography (EEG) in the EMU will be completed, epileptiform discharges (e.g., the number of spikes per 100 seconds, the number of seconds with spikes, and clinical seizures) will be counted before, during, and after music procedures. Heart rate variability and blood pressure will also be measured before, during, and after music stimuli. Participants' behavior changes will be recorded as a standard of care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Children with Epilepsy (Experimental): Children (age: 4- 17 years old) will participate in this study, and they will listen to Mozart K.448 (1st movement) and instrumental age-appropriate song with 10 minutes wash out in between, each lasting up to 9 minutes in the daytime (between 1-5 pm). The music stimuli will be randomly played in 2 to 7 days during the EMU stay (average 4 days). Music will be delivered via single-use earbuds.
  Interventions: Behavioral: Music Stimuli

INTERVENTIONS:
Behavioral: Music Stimuli — Nine-minute-long Mozart K.448 (1st movement) and instrumental age-appropriate songs will be played via single-use earbuds with 10 minutes wash-out in between music stimuli.

SUMMARY:
This research is being done to determine if Mozart music and/or age-appropriate music can reduce the frequency of seizures and epileptiform discharges.

DETAILED DESCRIPTION:
Several prospective studies have demonstrated the impact of Mozart's sonata for Two Pianos (K.448) on interictal epileptiform discharges and/or clinical seizure recurrence in children with epilepsy. While the exact mechanisms by which Mozart music has this effect are not yet established, there continues to be growing evidence demonstrating the positive effects on Mozart music upon seizure frequency and epileptiform discharges. Additional studies are needed to further elucidate the effect of Mozart music on epilepsy given the heterogeneity of protocols used in diverse clinical settings, with the goal of using these findings to drive potential therapy in the clinical setting.

Therefore, this study will explore if there are differences in epileptiform activity and clinical seizures between Mozart K.448, instrumental age-appropriate songs, and a patient's baseline activity during EMU stays. The children (age 4-17 yrs.) will listen to Mozart K.448 (1st movement) and instrumental age-appropriate songs with washout (10 minutes) in between, each lasting up to 9 minutes in the daytime. The music stimuli will be randomly played in 2 to 7 EMU stay days (average length of stay 4 days) and delivered via single-use earbuds. As per standard clinical care the investigators will monitor continuous video electroencephalography (EEG) in the epilepsy monitoring unit.

The frequency of epileptiform discharges (e.g., the number of spikes per 100 seconds, the number of seconds with spikes, and clinical seizures) will be counted before, during, and after music procedures. Heart rate variability and blood pressure will also be measured before, during, and after music stimuli to understand associations between physiological responses and epileptiform discharges to musical stimuli. Participants' behavior changes will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Children (age: 4 - 17 years old) who stay at Epilepsy Monitoring Units (EMU) up to 7 days may join.

Exclusion Criteria:

* Non-English Speaking

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2023-04-22 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in the frequency of epileptiform discharges (number of spikes) | Epilepsy Monitoring Units Stay (up to Day 7)
  The number of spikes in 100 seconds will be counted.
Change in the frequency of epileptiform discharges (number of seconds with spikes) | Epilepsy Monitoring Units Stay (up to Day 7)
  The number of seconds with spikes will be measured.

SECONDARY OUTCOMES:
Change in heart rate variability (HRV) | Epilepsy Monitoring Units Stay (up to Day 7)
  Heart rate variability (HRV) is the fluctuation in the time (ms) intervals between adjacent heartbeats.
Change in blood pressure variability (BPV) | Epilepsy Monitoring Units Stay (up to Day 7)
  The determinants of BPV are calculated for both systolic and diastolic blood pressure using "the indices standard deviation (SD), average real variability (ARV), and coefficient of variation (CV)" of all 3 measurement methods. The CV is obtained by dividing the SD by the average Blood Pressure (BP) level. The ARV is calculated as the average of the differences between consecutive BP measurements. SD, ARV and CV will be combined to report BPV. The unit of BPV is mmHg.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Kelley, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shaffer F, Ginsberg JP. An Overview of Heart Rate Variability Metrics and Norms. Front Public Health. 2017 Sep 28;5:258. doi: 10.3389/fpubh.2017.00258. eCollection 2017. PMID 29034226
- [Background] Abellan-Huerta J, Prieto-Valiente L, Montoro-Garcia S, Abellan-Aleman J, Soria-Arcos F. Correlation of Blood Pressure Variability as Measured By Clinic, Self-measurement at Home, and Ambulatory Blood Pressure Monitoring. Am J Hypertens. 2018 Feb 9;31(3):305-312. doi: 10.1093/ajh/hpx183. PMID 29040398
- [Background] Hernando-Requejo V. [Epilepsy, Mozart and his sonata K.448: is the <<Mozart effect>> therapeutic?]. Rev Neurol. 2018 May 1;66(9):308-314. Spanish. PMID 29696618
- [Background] Bedetti C, Principi M, Di Renzo A, Muti M, Frondizi D, Piccirilli M, D'Alessandro P, Marchiafava M, Baglioni A, Menna M, Gubbiotti M, Elisei S. The Effect of Mozart's Music in Severe Epilepsy: Functional and Morphological Features. Psychiatr Danub. 2019 Sep;31(Suppl 3):467-474. PMID 31488774